CLINICAL TRIAL: NCT03738722
Title: Positive Airway Pressure Under Apnoeic Oxygenation With Different Flow Rates
Brief Title: Positive Airway Pressure Under Apnoeic Oxygenation With Different Flow Rates in Nasal Cannula Therapy
Acronym: PAPUA-Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ID 2018-01834
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Apnoeic Oxygenation
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-flow-nasal-cannula-therapy (HFNCT) (Experimental): 100% Oxygen at 80 l/min with flow reductions of 20 l/min, jaw thrust, with opened and closed mouth, using different flow rates (80l/min, 60l/min, 40l/min, 20l/min, 1l/min) within each subject.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — HFNCT (high flow nasal cannula therapy) will be provided using OptiFlow by Fisher&Paykel.
  Other Names: High flow Oxygen

SUMMARY:
The main objective of this explorative observational study is to investigate the pressures in infraglottic airway and the pharynx provided by THRIVE , using flows ranging from 1l/min to 80 l/min, in patients hospitalized for elective surgical procedure; to investigate the correlation between airway pressure and nasal oxygen flow.

DETAILED DESCRIPTION:
Eligible adults with written informed consent will be monitored for general anaesthesia according standard operating procedure of the Bern University Hospital's anaesthesia department. Additional non-invasive monitoring for this study are transcutaneous measurement of carbon dioxide and oxygen (TCM 5®, Radiometer, Krefeld, Germany), NarcotrendTM ( Narcotrend-Group, Hannover, Germany)and thoracic electrical impedance tomography (EIT, PulmoVista® 500, Draeger, Luebeck, Germany).

Normal pre-oxygenation (until end expiratory carbon dioxide is > 90% or time > 3 minutes) will occur. Anaesthesia will be started using a target -controlled infusion system for Propofol and Remifentanil, using NarcotrendTM to measure depth of anaesthesia. All patients will receive a standard dose of neuromuscular blockage to facilitate airway management and total intravenous anaesthesia will be installed. Using the train of four measurement (TOF) full neuromuscular blockage with Rocuronium will be confirmed every 30 seconds. After administration of rocuronium, proper bag-mask ventilation will be confirmed.

Intratracheal pressure will be measured by 11 Fr. catheter (Cook Medical, Bloomington, IN, USA), connected to a CODAN Xtrans®-transducer (CODAN ARGUS Ag, Baar, Switzerland). A 11 Fr. catheter (Cook Medical, Bloomington, IN, USA) will be introduced oral in the trachea facilitated by video-laryngoscopy. To ensure patency of the upper airway jaw thrust via Esmarch manoeuvre will be applied and flexible bronchoscopy will confirm upper airway patency. Initially this 11 Fr. catheter will be positioned in the right main bronchus (2 cm below the carina). The first measurement will be performed with a randomized sequence of flow rates of 80, 60, 40, 20 or 1 l/min with opened and closed mouth. Each pressure measurement will be performed after a stable pressure plateau of 10 seconds will be observed. The catheter will then be retracted and the pressure quantification are performed with the same sequence, defined above, in different positions (50% of trachea length and pharyngeal pressures 10 cm from upper front teeth). The order of flow and mouth opening will be randomized.

The study intervention will end when all measurements are taken or upper airway patency cannot be ensured under direct endoscopy view. If one of the following criteria is met: peripheral oxygen saturation (SpO2) <92% or transcutaneous carbon dioxide (PtCO2) >80mmHg, immediately bag mask ventilation will be initiated, until normal values of SpO2 and PtCO2 are reached.

When any of the end points is reached, normal anesthesiologic care will be established as planned.

A safety interview will be conducted on the first post-operative day to evaluate injuries during airway management (e.g. bleeding, sore throat, hoarseness, lip injuries), pain, postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Written informed consent
* Undergoing elective surgery
* Requiring general anesthesia
* ASA 1-3 (American Society of Anesthesiologists)

Exclusion Criteria:

* Any Indication for fibre optic intubation
* Expected impossible mask ventilation
* Known coronary heart disease
* Known heart failure, NYHA classification( New York Heart Association ) ≥ 2
* Peripheral occlusive arterial disease, Fontaine ≥ 2b
* BMI > 30kg/m2 and BMI < 16kg/m2
* Hyperkalaemia (K > 5.5 mmol/l)
* Known COPD (Chronic obstructive pulmonary disease) Gold classification ≥ 2
* Known pulmonary arterial hypertension, systolic > 35mmHg
* Known obstructive sleep apnoea syndrome in need of therapy
* High risk of aspiration
* Increased intracranial pressure
* Intracranial surgery
* Limited knowledge of German language
* Absent power of judgement
* Pregnancy (pregnancy test before inclusion)
* Neuromuscular disorder
* Known or suspected cervical spine instability
* Nasal obstruction, impossibility of nasal ventilation (both sides patent)
* Allergies or contra-indications to one or more of the used anaesthesia agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Mean positive airway pressure during Apnoea (approx.10 min) with HFNCT (High-Flow-Nasal-Cannula-Therapy) | After induction of anaesthesia; Each pressure measurement (main bronchus,trachea, pharynx) will be performed after a stable pressure plateau of 10 sec. will be observed; until all measurements are taken or upper airway patency cannot be ensured
  Measurement of the mean positive airway pressure in cm H2O during apnoea time in the pharynx (10cm distal upper front teeth), in the trachea (50% length) and in the right main bronchus (2cm distal carina), with different flow-rates (80l/min, 60l/min, 40l/min, 20l/min, 1l/min), with opened and closed mouth

SECONDARY OUTCOMES:
Changes in ptcO2 and ptcCO2 in mmHg/min | After induction of anaesthesia, during apnoea period; until all pressure measurement (main bronchus,trachea, pharynx) are taken or upper airway patency cannot be ensured
  Transcutaneous measurement
Upper airway patency | After induction of anaesthesia, during apnoea period; until all pressure measurement (main bronchus,trachea, pharynx) are taken or upper airway patency cannot be ensured
  Flexible bronchoscopy will confirm upper airway patency: Open or closed
Changes in electrical impedance tomography. (EIT) | After induction of anaesthesia, during apnoea period; until all pressure measurement (main bronchus,trachea, pharynx) are taken or upper airway patency cannot be ensured
  EIT will be continuously measured using PulmoVista® 500 visualizing possible atelectasis formation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Principal Investigator — University hospital of Bern
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Riva T, Pedersen TH, Seiler S, Kasper N, Theiler L, Greif R, Kleine-Brueggeney M. Transnasal humidified rapid insufflation ventilatory exchange for oxygenation of children during apnoea: a prospective randomised controlled trial. Br J Anaesth. 2018 Mar;120(3):592-599. doi: 10.1016/j.bja.2017.12.017. Epub 2018 Jan 27. PMID 29452816
- [Background] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Background] Ritchie JE, Williams AB, Gerard C, Hockey H. Evaluation of a humidified nasal high-flow oxygen system, using oxygraphy, capnography and measurement of upper airway pressures. Anaesth Intensive Care. 2011 Nov;39(6):1103-10. doi: 10.1177/0310057X1103900620. PMID 22165366